CLINICAL TRIAL: NCT01861795
Title: An Oligo-center Observational Study to Collect Data in Preterm Neonates Born at or Above 27+0 Weeks of Gestational Age Who Are Sufficiently Stable on Non-Invasive Ventilatory Support
Brief Title: Observational Study in Preterm Neonates Who Are Sufficiently Stable on Non-Invasive Ventilatory Support
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: RS-7261-201-RD; U1111-1141-9396 (Registry Identifier: WHO)
Record Dates: First submitted 2013-04-26; First posted 2013-05-24 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Non-invasive Ventilatory Support; Infant Respiratory Distress Syndrome
Keywords: Drug therapy
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm Neonates: Preterm neonates born at or above 27+0 weeks of gestational age sufficiently stable on nasal continuous positive airway pressure (CPAP) will be treated by standard of care.
  Interventions: Other: Preterm Neonates

INTERVENTIONS:
Other: Preterm Neonates — Preterm Neonates

SUMMARY:
The purpose of this observational study is to collect data on vital signs, oxygen requirements and other data related to ventilator care in preterm neonates under standard of care treatment.

DETAILED DESCRIPTION:
The objective of this study is to collect data on vital signs, oxygen requirements and other data in preterm infants who are breathing stably on non-invasive ventilatory support. The data obtained during this study will be used to compare data obtained in a future study that will add a new medicinal product in combination with non-invasive ventilatory support to accelerate lung development in preterm infants.

The study will enroll approximately 40 patients. Participants will not be receiving any investigational medicinal product or device in this study.

All participants will have vital signs, oxygen requirements and other data collected continuously throughout the study.

This multi-centre trial will be conducted in Germany. The overall time to participate in this study is up to 10 weeks. Participants will be observed until they reach 36 weeks of gestational age or until they are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written, informed consent of both parents or legal guardian(s) obtained (on admission, prior to or after delivery).

  2. Preterm neonates born at or above 27+0 gestational weeks (GW) who are sufficiently stable on nasal continuous positive airway pressure (CPAP). Upper limit 36+0 GW.

  3. Participants' minimum weight at birth must be 800 g. Upper weight limit is 2500 g.

  4. CPAP-positive end-expiratory pressure (PEEP) must be ≥5 cm and ≤ 8 cm H2O. 5. Fraction of oxygen (O2) in ventilator outlet gas flow (FiO2) ≥ 30% to reach saturation goal (SpO2 between 88% and 96%) during the time period from B0 to T0.

Exclusion Criteria:

* 1. FiO2 > 50% to reach saturation goal (saturation of peripheral oxygen (SpO2) between 88% and 96%) during the time period from 30 minutes after birth (B0) to 45 minutes after birth (T0).

  2. Presence of severe respiratory distress syndrome (RDS) necessitating immediate intubation and surfactant rescue at entry into the study, or having necessitated surfactant rescue prior to entry into the study.

  3. Known life-threatening congenital anomaly or genetic syndrome. 4. Participation in an interventional study in parallel to this observational study.

Ages: 27 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates on non-invasive ventilatory support in a hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time and failure-adjusted Area Under the Curve (AUC) from Time 0 (T0) to 98 hours after T0 (T47) (AUCT0-T47adjusted) of fraction of inspired oxygen (FiO2) | Beginning of the Intensive observation phase (T0; approximately 45 minutes after birth) to 98 hours after T0
  Fraction of inspired oxygen (FiO2) is the amount of oxygen in the ventilator outlet gas flow.

SECONDARY OUTCOMES:
Time with optimal saturation of peripheral oxygen (SpO2) of 88% to 96% | T0 and at 0.25, 0.5, 0.75 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75 4, 4.25. 4.5, 4.74, 5, 5.25, 5.75, 6, 10, 14, 18, 22, 26, 30, 34, 38, 42, 46, 50, and 54 hours
  Saturation of peripheral oxygen is the amount of oxygen bound to hemoglobin in the blood expressed as a percentage of the maximal binding capacity. It will be measured with a pulse oximeter.
Continuous positive airway pressure (CPAP)-failure necessitating intubation and mechanical ventillation and/or surfactant instillation during observation period from T0 to 98 hours | T0 to 98 hours
  CPAP failure is reached when FiO2 ≥ 50% is need for more than 15 minutes to reach 90% saturation of peripheral oxygen (SpO2).
Percentage of participants requiring instillation of an approved surfactant preparation | Gestational week (GW) 36+6 days
Percentage of participants with bronchopulmonary dysplasia (BPD) at GW 36 | Gestational Week 36
  Bronchopulmonary dysplasia (BPD) is defined as a lung injury in preterm neonates resulting from oxygen toxicity and/or mechanical ventilation (elevated air pressure).
Respiratory rate over time | T0 to Gestational Week 36
Percentage of participants with a positive room-air challenge test at Gestational Week 36 | Gestational Week 36
  The room-air challenge test is defined as a weaning attempt allowing the participant to breath non-pressurized room air for 30 minutes. If a blood oxygen saturation of ≥90% is achieved during weaning, the weaning was successful and patients are considered to be free of bronchopulmonary dysplasia and need no further ventilation support.
Mortality rate | T0 to Gestational Week 36+6 days
Time under Continuous Positive Airway Pressure ventilatory support | T0 to Gestational Week 36+6 days
Time of additional oxygen demand (FiO2 > 21%) | T0 to Gestational Week 36+6 days
Time in neonatal intensive care unit (NICU) or intermediate care unit (IMCU) | T0 to Gestational Week 36+6 days
Time of intubation for mechanical ventilation | T0 to Gestational Week 36+6 days
Time on any ventilation support | T0 to Gestational Week 36+6 days
  Any ventilation support includes continuous positive airway pressure (CPAP), manual support and intubation.
Days in hospital | From T0 to Gestational Week 36+6 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (3):
- Germany (3):
  - Hanover
  - Lübeck
  - Nuremberg